CLINICAL TRIAL: NCT06973798
Title: The Study on the Effectiveness of [68Ga]Ga-HBED-CC-DiAsp PET/CT in Calculating Glomerular Filtration Rate and Predicting Residual Renal Function After Partial Nephrectomy
Brief Title: The Study on the Effectiveness of [68Ga]Ga-HBED-CC-DiAsp PET/CT in Calculating GFR and Predicting Residual Renal Function After Partial Nephrectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luo Yaping (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor-Investigator, Luo Yaping, Medical Doctor (M.D.), Chief Physician, Professor, Assistant Director, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HBED-CC; 2022-PUMCH-B-070 (Other Grant/Funding Number: Peking union medical college hospital)
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Kidney Neoplasms / Surgery; Glomerular Filtration Rate; Positron-Emission Tomography(PET)
Keywords: [68Ga]Ga-HBED-CC-DiAsp; PET/CT; glomerular filtration rate; partial nephrectomy
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients planned for partial nephrectomy due to renal tumors (Other)
  Interventions: Diagnostic Test: GFR will be measured using three methods at two weeks before surgery and four ± one week after surgery
- Subjects with varying levels of renal function and no history of renal tumors (Other)
  Interventions: Diagnostic Test: GFR will be measured using three methods: [68Ga]Ga-HBED-CC-DiAsp PET/CT, the Gates method, and the dual plasma sampling method with 99mTc-DTPA.

INTERVENTIONS:
Diagnostic Test: GFR will be measured using three methods at two weeks before surgery and four ± one week after surgery — GFR will be measured using three methods at two weeks before surgery and four ± one week after surgery
  Arms: Patients planned for partial nephrectomy due to renal tumors
Diagnostic Test: GFR will be measured using three methods: [68Ga]Ga-HBED-CC-DiAsp PET/CT, the Gates method, and the dual plasma sampling method with 99mTc-DTPA. — GFR will be measured using three methods: [68Ga]Ga-HBED-CC-DiAsp PET/CT, the Gates method, and the dual plasma sampling method with 99mTc-DTPA.
  Arms: Subjects with varying levels of renal function and no history of renal tumors

SUMMARY:
In subjects with different levels of renal function and no history of renal tumors, GFR is measured using [68Ga]Ga-HBED-CC-DiAsp PET/CT, the Gates method, and the 99mTc-DTPA dual plasma method. The consistency between the three methods is analyzed using intra-class correlation coefficient (ICC), concordance correlation coefficient (CCC), and Bland-Altman analysis.

In patients scheduled for partial nephrectomy due to renal tumors, GFR is measured using the three methods within 2 weeks before surgery and 4±1 weeks post-surgery. The percentage of postoperative residual renal function (postoperative GFR/preoperative GFR × 100%, hereafter referred to as RRF%) is calculated for each method. By comparing and overlaying preoperative and postoperative PET/CT images, the resected renal area can be delineated on the preoperative PET/CT image. Based on the preoperative PET/CT and the delineated surgical area, a predictive value for postoperative GFR is calculated to obtain the predicted RRF%. A consistency analysis is then performed between the predicted RRF% and the actual RRF% measured by the three methods, using ICC, CCC, and Bland-Altman analysis to evaluate the efficacy of [68Ga]Ga-HBED-CC-DiAsp PET/CT in predicting residual renal function after partial nephrectomy.

DETAILED DESCRIPTION:
[68Ga]Ga-HBED-CC-DiAsp PET/CT Imaging: After intravenous injection of [68Ga]Ga-HBED-CC-DiAsp, a Scout scan, low-dose CT scan, and a 30-minute dynamic PET scan are performed sequentially. The functional renal cortex is delineated in the first PET frame showing the radiotracer filling the renal cortex. A functional renal cortex radioactivity concentration function is constructed based on a compartment model with GFR as a parameter and time as an independent variable. This function is then fitted to the time-activity curve (TAC) of the functional renal cortex to obtain the GFR value.

Gates Method and 99mTc-DTPA Dual Plasma Method: After intravenous injection of 99mTc-DTPA, renal blood flow functional imaging is performed immediately, collecting time-activity curves from both renal areas. GFR is calculated based on the percentage (%ID) of bilateral renal radiotracer uptake relative to the injected dose. Blood samples of 10 ml are collected from the contralateral forearm at 1 hour and 2 hours post-injection, and GFR is calculated using the dual plasma method.

In subjects with different levels of renal function and no history of renal tumors, GFR is measured using [68Ga]Ga-HBED-CC-DiAsp PET/CT, the Gates method, and the 99mTc-DTPA dual plasma method. The consistency between the three methods is analyzed using intra-class correlation coefficient (ICC), concordance correlation coefficient (CCC), and Bland-Altman analysis.

In patients scheduled for partial nephrectomy due to renal tumors, GFR is measured using the three methods within 2 weeks before surgery and 4±1 weeks post-surgery. The percentage of postoperative residual renal function (postoperative GFR/preoperative GFR × 100%, hereafter referred to as RRF%) is calculated for each method. By comparing and overlaying preoperative and postoperative PET/CT images, the resected renal area can be delineated on the preoperative PET/CT image. Based on the preoperative PET/CT and the delineated surgical area, a predictive value for postoperative GFR is calculated to obtain the predicted RRF%. A consistency analysis is then performed between the predicted RRF% and the actual RRF% measured by the three methods, using ICC, CCC, and Bland-Altman analysis to evaluate the efficacy of [68Ga]Ga-HBED-CC-DiAsp PET/CT in predicting residual renal function after partial nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Written informed consent obtained.

Exclusion Criteria:

* Patients with claustrophobia or fear of radiation;
* Women who are planning to conceive, pregnant, or breastfeeding;
* Patients unable to lie flat for 30 minutes;
* Patients or family members who cannot understand the conditions and objectives of the study, or who refuse to participate.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
glomerular filtration rate | From enrollment to the end of examination at 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Due to patient privacy regulations and institutional policies, individual participant data (IPD) from this study will not be publicly available. The data contain sensitive clinical and genetic information that could compromise participant confidentiality. Additionally, Chinese data protection laws and hospital ethical guidelines restrict the open sharing of identifiable medical data.
  However, aggregated results (e.g., group-level imaging findings, statistical analyses) will be published in peer-reviewed journals. Researchers may request limited, anonymized datasets for collaborative purposes, subject to approval by the Peking Union Medical College Hospital (PUMCH) Ethics Committee and compliance with data transfer agreements.

REFERENCES:
- [Background] Shi S, Zhang L, Wu Z, Zhang A, Hong H, Choi SR, Zhu L, Kung HF. [68Ga]Ga-HBED-CC-DiAsp: A new renal function imaging agent. Nucl Med Biol. 2020 Mar-Apr;82-83:17-24. doi: 10.1016/j.nucmedbio.2019.12.005. Epub 2019 Dec 16. PMID 31869735
- [Background] Rathi N, Attawettayanon W, Kazama A, Yasuda Y, Munoz-Lopez C, Lewis K, Maina E, Wood A, Palacios DA, Li J, Abdallah N, Weight CJ, Eltemamy M, Krishnamurthi V, Abouassaly R, Campbell SC. Practical Prediction of New Baseline Renal Function After Partial Nephrectomy. Ann Surg Oncol. 2024 Feb;31(2):1402-1409. doi: 10.1245/s10434-023-14540-x. Epub 2023 Nov 25. PMID 38006535
- [Background] Murray AW, Barnfield MC, Waller ML, Telford T, Peters AM. Assessment of glomerular filtration rate measurement with plasma sampling: a technical review. J Nucl Med Technol. 2013 Jun;41(2):67-75. doi: 10.2967/jnmt.113.121004. Epub 2013 May 8. PMID 23658207
- [Background] Hofman MS, Hicks RJ. Gallium-68 EDTA PET/CT for Renal Imaging. Semin Nucl Med. 2016 Sep;46(5):448-61. doi: 10.1053/j.semnuclmed.2016.04.002. PMID 27553470
- [Background] Hofman M, Binns D, Johnston V, Siva S, Thompson M, Eu P, Collins M, Hicks RJ. 68Ga-EDTA PET/CT imaging and plasma clearance for glomerular filtration rate quantification: comparison to conventional 51Cr-EDTA. J Nucl Med. 2015 Mar;56(3):405-9. doi: 10.2967/jnumed.114.147843. Epub 2015 Feb 12. PMID 25678493
- [Background] Gates GF. Computation of glomerular filtration rate with Tc-99m DTPA: an in-house computer program. J Nucl Med. 1984 May;25(5):613-8. PMID 6374072